CLINICAL TRIAL: NCT01405053
Title: A Multicenter, Randomized, Controlled, Open-label Study to Evaluate the Cognitive Development Effects and Safety, and Pharmacokinetics of Adjunctive Rufinamide Treatment in Pediatric Subjects 1 to Less Than 4 Years of Age With Inadequately Controlled Lennox-Gastaut Syndrome
Brief Title: Study of Rufinamide in Pediatric Subjects 1 to Less Than 4 Years of Age With Lennox-Gastaut Syndrome Inadequately Controlled With Other Anti-epileptic Drugs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2080-G000-303
Expanded Access: Available
Record Dates: First submitted 2011-07-27; First posted 2011-07-29 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2016-02

CONDITIONS: Lennox-Gastaut Syndrome
Keywords: Central Nervous System
MeSH Terms: conditions — Lennox Gastaut Syndrome | interventions — rufinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rufinamide (Active Comparator)
  Interventions: Drug: Rufinamide
- Any other approved AED (Active Comparator)
  Interventions: Drug: Any other approved Antiepileptic Drug

INTERVENTIONS:
Drug: Rufinamide — Rufinamide up to 45 mg/kg/day, in 2 divided doses, administered as oral suspension (40 mg/mL) as an add-on to the subject's existing regimen of 1-3 antiepileptic drugs (AEDs)
  Arms: Rufinamide
Drug: Any other approved Antiepileptic Drug — Any other approved AED: any other approved AED of the investigator's choice as an add-on to the subject's existing regimen of 1-3 anti-epileptic drugs (AEDs)
  Arms: Any other approved AED

SUMMARY:
This study was designed to evaluate the cognitive effect, safety, and pharmacokinetics (PK) of rufinamide on Lennox-Gastaut Syndrome (LGS) inadequately controlled in pediatric participants already taking other anti-epileptic drugs.

ELIGIBILITY:
Key Inclusion:

1. Clinical diagnosis of LGS, which might include the presence of a slow background electroencephalogram (EEG) rhythm, slow spikes-waves pattern (less than 3 Hz), the presence of polyspikes; care should be taken not to include benign myoclonic epilepsy of infancy, atypical benign partial epilepsy (pseudo-Lennox syndrome), or continuous spike-waves of slow sleep (CSWS).
2. On a fixed and documented dose of one to three concomitant regionally approved antiepileptic drugs (AEDs) for a minimum of 4 weeks prior to randomization with an inadequate response to treatment.
3. Consistent seizure documentation (i.e., no uncertainty of the presence of seizures) during the pre-randomization phase.

Key Exclusion:

1. Familial short QT syndrome
2. Prior treatment with rufinamide within 30 days of baseline visit or discontinuation of rufinamide treatment due to safety issues related to rufinamide

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2011-06-16 (Actual); Primary Completion 2015-11-02 (Actual); Study Completion 2015-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Arzimanoglou Arzimanoglou, Principal Investigator — Hopital Femme-Mere-Enfant Service D'Epilepsie -5eme etage 59 Boulevard Pinel Bron, France
Locations (47):
- United States (22):
  - San Diego, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Gulf Breeze, Florida
  - Miami, Florida
  - Tampa, Florida
  - Wellington, Florida
  - Augusta, Georgia
  - Chicago, Illinois
  - Lexington, Kentucky
  - Shreveport, Louisiana
  - Lebanon, New Hampshire
  - Gibbsboro, New Jersey
  - Rochester, New York
  - Akron, Ohio
  - Akson, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Austin, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
- Canada (4):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Toronto, Ontario
  - Saskatoon
- France (3):
  - Bron
  - Marseille
  - Paris
- Greece (4):
  - Ambelokipi Athens
  - Pátrai
  - Pendeli Athens
  - Thessaloniki
- Italy (7):
  - Mantova, MN
  - Calambrone, PI
  - Pisa, PI
  - Pavia, PV
  - Mantova
  - Roma
  - Salerno
- Poland (6):
  - Elblag
  - Gdansk
  - Kielce
  - Poznan
  - Rzeszów
  - Warsaw
- Cape Town, South Africa

REFERENCES:
- [Derived] Brigo F, Jones K, Eltze C, Matricardi S. Anti-seizure medications for Lennox-Gastaut syndrome. Cochrane Database Syst Rev. 2021 Apr 7;4(4):CD003277. doi: 10.1002/14651858.CD003277.pub4. PMID 33825230
- [Derived] Auvin S, Williams B, McMurray R, Kumar D, Perdomo C, Malhotra M. Novel seizure outcomes in patients with Lennox-Gastaut syndrome: Post hoc analysis of seizure-free days in rufinamide Study 303. Epilepsia Open. 2019 Mar 13;4(2):275-280. doi: 10.1002/epi4.12314. eCollection 2019 Jun. PMID 31168494
- [Derived] Arzimanoglou A, Ferreira J, Satlin A, Olhaye O, Kumar D, Dhadda S, Bibbiani F. Evaluation of long-term safety, tolerability, and behavioral outcomes with adjunctive rufinamide in pediatric patients (>/=1 to <4 years old) with Lennox-Gastaut syndrome: Final results from randomized study 303. Eur J Paediatr Neurol. 2019 Jan;23(1):126-135. doi: 10.1016/j.ejpn.2018.09.010. Epub 2018 Sep 27. PMID 30309816
- [Derived] Arzimanoglou A, Ferreira JA, Satlin A, Mendes S, Williams B, Critchley D, Schuck E, Hussein Z, Kumar D, Dhadda S, Bibbiani F. Safety and pharmacokinetic profile of rufinamide in pediatric patients aged less than 4 years with Lennox-Gastaut syndrome: An interim analysis from a multicenter, randomized, active-controlled, open-label study. Eur J Paediatr Neurol. 2016 May;20(3):393-402. doi: 10.1016/j.ejpn.2015.12.015. Epub 2016 Jan 11. PMID 26805435

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 19 investigative sites in the United States, Canada, France, Greece, Italy, and Poland from 16 June 2011 to 02 November 2015.
Pre-assignment Details: A total of 43 participants were screened, out of which 37 participants were randomized and treated in the study.
Groups:
- Rufinamide: Participants received rufinamide oral suspension as an add-on therapy to the participant's existing regimen of 1 to 3 Antiepileptic Drugs (AEDs). Participants underwent a 2 week Titration Period during which rufinamide dose was increased from 10 milligram per kilogram per day (mg/kg/day) in increments of 10 mg/kg/day every 3 days to 40 mg/kg/day and thereafter in increments of 5 mg/kg/day to the target maintenance dose of 45 mg/kg/day (all daily treatments were to be administered in 2 equally divided doses). Rufinamide dose reached at the end of the Titration period were to be maintained the same throughout the 104-week Maintenance Period. At the end of Maintenance Period, rufinamide dose should be tapered (as needed) over a period of 2 weeks.
- Any Other Approved Antiepileptic Drug: Participants received any other approved AEDs of the investigator's choice, dosed according to the investigator's usual practice, added to the participant's existing regimen of 1 to 3 AEDs. At the end of Maintenance Period, the AED comparator would be discontinued according to the investigator's usual practice.
Period: Overall Study
Arm/Group | Rufinamide | Any Other Approved Antiepileptic Drug
Started | 25 | 12
Completed | 15 | 4
Not Completed | 10 | 8
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Participant choice | 2 | 1
Not completed — Inadequate therapeutic effect | 2 | 1
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all enrolled participants who received at least 1 dose of rufinamide or any other approved add-on AED of the investigator's choice and had at least 1 postdose safety assessment.
Groups:
- Rufinamide: Participants received rufinamide oral suspension as an add-on therapy to the participant's existing regimen of 1 to 3 AEDs. Participants underwent a 2 week Titration Period during which rufinamide dose was increased from 10 mg/kg/day in increments of 10 mg/kg/day every 3 days to 40 mg/kg/day and thereafter in increments of 5 mg/kg/day to the target maintenance dose of 45 mg/kg/day (all daily treatments were to be administered in 2 equally divided doses). Rufinamide dose reached at the end of the Titration period were to be maintained the same throughout the 104-week Maintenance Period. At the end of Maintenance Period, rufinamide dose should be tapered (as needed) over a period of 2 weeks.
- Total: Total of all reporting groups
Arm/Group | Rufinamide | Any Other Approved Antiepileptic Drug | Total
Number analyzed (Participants) | 25 | 12 | 37
Age, Continuous [Mean (Standard Deviation); unit: months] | 28.3 (9.99) | 29.8 (9.85) | 28.8 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 13
  Male | 14 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Child Behavior Checklist (CBCL) Total Problem T-scores at the End of 2-year Treatment Period
Description: CBCL: 99-item questionnaire measures specific behavioral problems or developmental delays, answered by a parent/legal guardian or suitable caregiver. Each item were rated using 3-point scale (0=Not True, 1=Somewhat/Sometimes True, 2=Very True/ Often True) to indicate how often or typical the behavior was. The 99 items were combined to yield scores for 8 problem area scales (emotionally reactive, anxious/depressed, somatic complaints, withdrawn, sleep problems, attention problems, aggressive behavior, and other problems) and 3 summary scores (internalizing, externalizing, and total problems). Total Problem score was sum of all the problem areas plus 1 additional item, ranging from 0 to 198. Total raw scores are converted to t-scores with mean of 50 and standard deviation (SD) of 10. T-scores were standardized test scores that indicate same degree of elevation in problems relative to the normative sample of peers. Higher scores were indicative of more problems.
Time Frame: End of Treatment Period (up to approximately Week 106)
Population: The full analysis set for primary efficacy variable included randomized participants who received rufinamide or any other approved add-on AED of the investigator's choice and had baseline and at least 1 postdose cognition measurement. Participants who were evaluable for this outcome measure at given time period were included for assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rufinamide | Any Other Approved Antiepileptic Drug
Number analyzed (Participants) | 15 | 4
score on a scale | 55.7 (15.81) | 54.8 (4.50)
Statistical Analysis 1: Comparison: Rufinamide vs Any Other Approved Antiepileptic Drug; The primary statistical model for comparing the 2 treatment groups was an analysis of covariance (ANCOVA) mixed model for repeated measures with baseline score, age, and sex as covariates, and treatment, week, and treatment by week interaction as factors; Test type: Superiority; p = 0.6928, ANCOVA; LS Mean difference = 2.601, 95% CI 2-sided [-10.5 to 15.7], Standard Error of Mean 6.558

2. Primary Outcome: Change From Baseline in CBCL Total Problem T-Scores at End of 2-year Treatment Period
Description: as for outcome 1
Time Frame: Baseline and End of Treatment Period (up to approximately Week 106)
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rufinamide | Any Other Approved Antiepileptic Drug
Number analyzed (Participants) | 24 | 9
score on a scale
  Baseline: number analyzed (Participants) | 24 | 8
  Baseline | 56.6 (11.27) | 62.8 (13.07)
  Change at Week 106: number analyzed (Participants) | 15 | 3
  Change at Week 106 | -0.3 (15.72) | -6.7 (0.58)

3. Other Pre Specified Outcome: Time to Withdrawal From Treatment Due to an Adverse Event or Lack of Efficacy
Description: Withdrawal from either rufinamide or other AED was due to the occurrence of an adverse event or for lack of efficacy. Data was obtained till Week 106 and was extrapolated using Kaplan-Meier method to determine the overall survival time (in weeks) to withdrawal from treatment (excluding taper) due to an adverse event or lack efficacy.
Time Frame: Baseline up to the End of the Treatment Period (up to approximately Week 106)
Population: The full analysis set for other efficacy variable included randomized participants who received rufinamide or any other add-on AED of the investigator's choice and had a baseline efficacy assessment and at least 1 post baseline efficacy assessment. Participants who were evaluable at a given time point were included for this assessment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Rufinamide | Any Other Approved Antiepileptic Drug
Number analyzed (Participants) | 2 | 2
weeks | 142.0 [NA to NA] — NA: Lower and upper limits of 95% Confidence Interval could not be calculated since insufficient number of participants had withdrawal from treatment due to adverse event or lack of efficacy. | 28.0 [17.7 to NA] — NA: Lower and upper limits of 95% Confidence Interval could not be calculated since insufficient number of participants had withdrawal from treatment due to adverse event or lack of efficacy.

4. Other Pre Specified Outcome: Percent Change in Total Seizure Frequency Per 28 Days
Description: The frequency per 28 days was defined as (S/D)*28 where, S was equal to the sum of the seizures reported in the participant seizure diary during the specified time interval and D was equal to the number of days with non-missing data in the participant seizure diary for the specified study phase. The number of seizures was assessed and recorded by the participant's parent(s)/caregiver(s) in the participant seizure diary.
Time Frame: Baseline up to End of the Treatment Period (up to approximately Week 106)
Population: The full analysis set for other efficacy variable included randomized participants who received rufinamide or any other add-on AED of the investigator's choice and had a baseline efficacy assessment and at least 1 postbaseline efficacy assessment. Participants evaluable for this outcome measure at given time period were included for assessment.
Measure: Median (Full Range); unit: percent change in seizure frequency
Arm/Group | Rufinamide | Any Other Approved Antiepileptic Drug
Number analyzed (Participants) | 24 | 8
percent change in seizure frequency | -7.05 [-79.2 to 3644.1] | -20.15 [-83.3 to 143.1]

5. Other Pre Specified Outcome: Percent Change in Seizure Frequency by Individual Seizure Type Per 28 Days
Description: as for outcome 4
Time Frame: Baseline up to End of Treatment Period (up to approximately Week 106)
Population: as for outcome 4
Measure: Median (Full Range); unit: percent change in seizure frequency
Arm/Group | Rufinamide | Any Other Approved Antiepileptic Drug
Number analyzed (Participants) | 24 | 9
percent change in seizure frequency
  Partial seizures: number analyzed (Participants) | 12 | 2
  Partial seizures | -39.8 [-100.0 to 52281.9] | -57.65 [-98.1 to -17.2]
  Absence seizures: number analyzed (Participants) | 11 | 5
  Absence seizures | -23.6 [-100.0 to 86.8] | -49.70 [-98.9 to 1846.7]
  Atypical absence seizures: number analyzed (Participants) | 14 | 4
  Atypical absence seizures | -70.95 [-100.0 to 16825.4] | 4.90 [-90.9 to 1189.7]
  Myoclonic seizures: number analyzed (Participants) | 13 | 4
  Myoclonic seizures | -24.60 [-73.3 to 11462.4] | -27.90 [-60.9 to 130.2]
  Clonic seizures: number analyzed (Participants) | 6 | 2
  Clonic seizures | -60.85 [-100.0 to 140.4] | -48.35 [-54.2 to -42.5]
  Tonic-atonic seizures: number analyzed (Participants) | 17 | 4
  Tonic-atonic seizures | -35.20 [-100.0 to 1250.6] | -31.80 [-81.9 to -4.0]
  Primary generalized tonic-clonic seizures: number analyzed (Participants) | 7 | 1
  Primary generalized tonic-clonic seizures | -97.80 [-100.0 to 37.6] | -96.60 [-96.6 to -96.6]
  Other seizures: number analyzed (Participants) | 10 | 3
  Other seizures | -90.65 [-100.0 to 183.8] | -100.00 [-100.0 to -54.0]

6. Other Pre Specified Outcome: Incidence of Worsening of Seizures
Description: Worsening of seizures was summarized by the incidence of participants with doubling in total seizure frequency, doubling in frequency of major seizures (generalized tonic-clonic, drop attacks), or occurrence of new seizure type during each successive 3 to 4 month visit interval of the Maintenance Period relative to baseline.
Time Frame: Baseline up to End of Treatment Period (up to approximately Week 106)
Population: The full analysis set for other efficacy variable included randomized participants who received rufinamide or any other add-on AED of the investigator's choice and had a baseline efficacy assessment and at least 1 postbaseline efficacy assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Rufinamide | Any Other Approved Antiepileptic Drug
Number analyzed (Participants) | 24 | 9
Participants
  Doubling in total seizure frequency | 4 | 1
  Doubling in frequency of major seizures | 5 | 1
  Occurrence of a new seizure type | 0 | 0

7. Other Pre Specified Outcome: Change From Baseline in CBCL Sub Scores at Week 106
Description: CBCL: 99-item questionnaire, measures behavioral problems/developmental delays, answered by parent/guardian/caregiver. Each item rated on 3-point scale (0=Not True,1=Somewhat/Sometimes True, 2=Very/Often True). 99 items were combined to give scores for 8 problem area scales, where 1 for each 8 syndrome (emotionally reactive, anxious/depressed, somatic, withdrawn, sleep, attention, aggressive behavior, and other problems) were calculated, range: 0 (normal) to 16 (clinical behavior) and 3 summary scores (internalizing, externalizing, and total problems). All 3 summary scores reported scaled to T-scores. Total Problem score was sum of all the problem areas plus 1 additional item, ranging from 0 to 198. Total raw score were converted to t-scores with mean of 50 and SD of 10. T-scores were standardized test scores that indicate same degree of elevation in problems relative to normative sample of peers. Higher scores were indicative of more problems.
Time Frame: Baseline and Week 106
Population: The full analysis set for other efficacy variable included randomized participants who received rufinamide or any other approved add-on AED of the investigator's choice and had a baseline efficacy and at least 1 postbaseline efficacy assessment. Participants evaluable for this outcome measure at given time period were included for assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rufinamide | Any Other Approved Antiepileptic Drug
Number analyzed (Participants) | 24 | 9
score on a scale
  Baseline: Total emotional reactive scores: number analyzed (Participants) | 24 | 8
  Baseline: Total emotional reactive scores | 59.0 (8.13) | 60.9 (8.64)
  Change at Week 106:Total emotional reactive scores: number analyzed (Participants) | 15 | 3
  Change at Week 106:Total emotional reactive scores | -1.1 (9.30) | -1.3 (6.11)
  Baseline: Total anxious/depression scores: number analyzed (Participants) | 24 | 8
  Baseline: Total anxious/depression scores | 56.4 (7.48) | 54.6 (6.67)
  Change at Week 106:Total anxious/depression scores: number analyzed (Participants) | 15 | 3
  Change at Week 106:Total anxious/depression scores | 0.5 (8.87) | 0.7 (1.15)
  Baseline: Total Somatic Complaints Scores: number analyzed (Participants) | 24 | 8
  Baseline: Total Somatic Complaints Scores | 59.4 (8.13) | 54.9 (4.70)
  Change at Week 106:Total Somatic Complaints Scores: number analyzed (Participants) | 15 | 3
  Change at Week 106:Total Somatic Complaints Scores | 0.1 (11.24) | -1.7 (2.89)
  Baseline: Total withdrawn scores: number analyzed (Participants) | 24 | 8
  Baseline: Total withdrawn scores | 71.5 (11.72) | 72.1 (11.03)
  Change at Week 106:Total withdrawn scores: number analyzed (Participants) | 15 | 3
  Change at Week 106:Total withdrawn scores | -2.2 (13.22) | -7.0 (9.54)
  Baseline: Total Sleep Problems Scores: number analyzed (Participants) | 24 | 8
  Baseline: Total Sleep Problems Scores | 57.8 (10.72) | 62.4 (8.57)
  Change at Week 106:Total sleep problem scores: number analyzed (Participants) | 15 | 3
  Change at Week 106:Total sleep problem scores | -1.9 (12.30) | -5.7 (7.57)
  Baseline: Total attention problems scores: number analyzed (Participants) | 24 | 8
  Baseline: Total attention problems scores | 59.3 (9.17) | 65.9 (10.72)
  Change at Week 106:Total attention problems scores: number analyzed (Participants) | 15 | 3
  Change at Week 106:Total attention problems scores | -1.1 (4.65) | -7.7 (2.52)
  Baseline: Total Aggressive Behavior Scores: number analyzed (Participants) | 24 | 8
  Baseline: Total Aggressive Behavior Scores | 52.5 (5.01) | 58.6 (12.07)
  Change at Week106:Total aggressive behavior scores: number analyzed (Participants) | 15 | 3
  Change at Week106:Total aggressive behavior scores | 3.2 (6.26) | -0.3 (2.89)
  Baseline: Total internalizing scores: number analyzed (Participants) | 24 | 8
  Baseline: Total internalizing scores | 61.6 (10.78) | 60.6 (9.71)
  Change at Week 106:Total internalizing scores: number analyzed (Participants) | 15 | 3
  Change at Week 106:Total internalizing scores | -1.5 (13.73) | -2.7 (1.53)
  Baseline: Total externalizing scores: number analyzed (Participants) | 24 | 8
  Baseline: Total externalizing scores | 47.5 (11.22) | 58.1 (15.92)
  Change at Week 106:Total externalizing scores: number analyzed (Participants) | 15 | 3
  Change at Week 106:Total externalizing scores | 4.7 (10.07) | -3.7 (3.51)

8. Other Pre Specified Outcome: Change From Baseline in Language Development Survey (LDS) Scores During Maintenance Period
Description: LDS, a caregiver-administered survey consisted of 8-item questionnaire and vocabulary list of 310 words organized within 14 semantic categories. List contained high frequency words (e.g. more), less common words (e.g. hamburger), and lexical chunks (e.g. Sesame Street). Average LDS score, calculated by dividing total number of words across all valid phrases by number of phrases with greater than (>) 0words; for participants with no words, average was 0. This value was compared to standardized chart to obtain percentile rating. LDS provided 2 scores: average phrase length (number of words/phrase) and number of endorsed vocabulary words. LDS phrase length was categorized into delay (less than or equal to [<=] 20th percentile) and no delay (>20th percentile). LDS vocabulary was categorized into delay(<=15th percentile)and no delay(>15th percentile). Both raw scores were used to provide 2 normative scores based on child's age in months. Higher scores indicated better language development.
Time Frame: Baseline, Weeks 24, 56, 88, and 106
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Rufinamide | Any Other Approved Antiepileptic Drug
Number analyzed (Participants) | 24 | 9
words
  Baseline: LDS average phrase length | 0.3 (0.87) | 0 (0.00)
  Change at Week 24: LDS average phrase length: number analyzed (Participants) | 23 | 8
  Change at Week 24: LDS average phrase length | 0.2 (1.11) | 0.7 (1.28)
  Change at Week 56: LDS average phrase length: number analyzed (Participants) | 21 | 7
  Change at Week 56: LDS average phrase length | 0.1 (1.02) | 0.0 (0.00)
  Change at Week 88: LDS average phrase length: number analyzed (Participants) | 18 | 4
  Change at Week 88: LDS average phrase length | 0.1 (1.03) | 0.0 (0.00)
  Change at Week 106: LDS average phrase length: number analyzed (Participants) | 16 | 4
  Change at Week 106: LDS average phrase length | 0.4 (1.12) | 0.0 (0.00)
  Baseline:LDS Vocabulary Score | 10.4 (37.72) | 0.6 (1.67)
  Change at Week 24:LDS Vocabulary Score: number analyzed (Participants) | 23 | 8
  Change at Week 24:LDS Vocabulary Score | 7.1 (21.55) | 4.8 (8.22)
  Change at Week 56:LDS Vocabulary Score: number analyzed (Participants) | 21 | 7
  Change at Week 56:LDS Vocabulary Score | 17.9 (39.24) | -0.40 (2.15)
  Change at Week 88:LDS Vocabulary Score: number analyzed (Participants) | 18 | 4
  Change at Week 88:LDS Vocabulary Score | 25.4 (49.87) | 0.0 (0.00)
  Change at Week 106:LDS Vocabulary Score: number analyzed (Participants) | 16 | 4
  Change at Week 106:LDS Vocabulary Score | 39.6 (75.62) | 1.0 (2.00)

9. Other Pre Specified Outcome: Change From Baseline in Total Score of Quality of Life in Childhood Epilepsy (QoLCE) Scale
Description: The QoLCE was a 76-item questionnaire designed specifically to measure quality of life in children with epilepsy. QOLCE consists of 16 quality of life subscales (14 multi-item and 2 single item). Each subscales had number of items or questions with responses as excellent, very good, good, fair, and poor. They were changed to 1, 2, 3, 4, and 5 as per instructions. Then changed on a scale of 100, where 1 is equal to (=) 0, 2=25, 3=50, 4=75, and 5=100. Items corresponding to each subscale were marked and there mean score was score of that subscale. The form was completed by a parent or caregiver who interacted with the child on a consistent, daily basis and took about 20 to 30 minutes to complete. The higher the score, the better the child's quality of life.
Time Frame: Baseline and Week 106
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rufinamide | Any Other Approved Antiepileptic Drug
Number analyzed (Participants) | 24 | 9
score on a scale
  Baseline | 50.4 (10.05) | 49.6 (7.88)
  Week 106: number analyzed (Participants) | 15 | 4
  Week 106 | -1.3 (8.49) | 1.5 (1.00)

10. Other Pre Specified Outcome: Change From Baseline in Sub-scores in QoLCE
Description: The QoLCE was a 76-item questionnaire designed specifically to measure quality of life in children with epilepsy. QOLCE consists of 16 quality of life subscales (14 multi-item and 2 single item). Each subscales had number of items or questions with responses as excellent, very good, good, fair, and poor. They were changed to 1, 2, 3, 4, and 5 as per instructions. Then changed on a scale of 100, where 1=0, 2=25, 3=50, 4=75, and 5=100. Items corresponding to each subscale were marked and there mean score was score of that subscale. The form was completed by a parent or caregiver who interacted with the child on a consistent, daily basis and took about 20 to 30 minutes to complete. The higher the score, the better the child's quality of life.
Time Frame: Baseline and Week 106
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rufinamide | Any Other Approved Antiepileptic Drug
Number analyzed (Participants) | 24 | 9
score on a scale
  Baseline: Physical restriction | 50.1 (10.33) | 49.9 (8.23)
  Change at Week 106: Physical restriction: number analyzed (Participants) | 15 | 4
  Change at Week 106: Physical restriction | -1.0 (7.51) | -6.8 (7.32)
  Baseline: Energy/Fatigue | 51.6 (10.48) | 44.3 (4.55)
  Change at Week 106: Energy/Fatigue: number analyzed (Participants) | 15 | 4
  Change at Week 106: Energy/Fatigue | -3.1 (12.22) | 2.8 (4.11)
  Baseline: Attention/Concentration | 49.9 (10.14) | 51.1 (9.05)
  Change at Week 106:Attention/Concentration: number analyzed (Participants) | 15 | 4
  Change at Week 106:Attention/Concentration | -2.1 (7.31) | 2.5 (6.24)
  Baseline: Memory | 50.2 (9.54) | 52.6 (6.57)
  Change at Week 106: Memory: number analyzed (Participants) | 15 | 4
  Change at Week 106: Memory | -0.5 (12.18) | 0.5 (1.00)
  Baseline: Language | 49.8 (10.42) | 53.1 (4.43)
  Change at Week 106: Language: number analyzed (Participants) | 15 | 4
  Change at Week 106: Language | -0.5 (9.63) | -0.5 (11.56)
  Baseline: Other cognitive | 48.6 (10.32) | 53.1 (7.54)
  Change at Week 106: Other cognitive: number analyzed (Participants) | 15 | 4
  Change at Week 106: Other cognitive | 0.3 (6.19) | -1.0 (4.00)
  Baseline: Depression | 51.2 (9.27) | 45.3 (10.59)
  Change at Week 106: Depression: number analyzed (Participants) | 15 | 4
  Change at Week 106: Depression | -2.6 (11.64) | 2.3 (8.62)
  Baseline: Anxiety | 50.1 (10.27) | 48.5 (12.29)
  Change at Week 106: Anxiety: number analyzed (Participants) | 15 | 4
  Change at Week 106: Anxiety | -0.1 (12.12) | 1.3 (6.90)
  Baseline: Control/Helplessness | 50.7 (9.31) | 47.8 (12.27)
  Change at Week 106: Control/Helplessness: number analyzed (Participants) | 15 | 4
  Change at Week 106: Control/Helplessness | 0.2 (10.90) | 3.0 (11.52)
  Baseline: Self-esteem | 50.1 (10.18) | 50.5 (10.98)
  Change at Week 106: Self-esteem: number analyzed (Participants) | 15 | 4
  Change at Week 106: Self-esteem | -1.3 (9.48) | -6.0 (8.08)
  Baseline: Social interactions | 49.9 (10.56) | 50.5 (8.48)
  Change at Week 106: Social interactions: number analyzed (Participants) | 15 | 4
  Change at Week 106: Social interactions | -1.5 (11.64) | 4.0 (5.89)
  Baseline: Social activities | 50.5 (10.50) | 46.6 (3.96)
  Change at Week 106: Social activities: number analyzed (Participants) | 15 | 4
  Change at Week 106: Social activities | 0.9 (11.30) | 3.5 (3.70)
  Baseline: Stigma | 48.9 (11.06) | 50.7 (8.07)
  Change at Week 106: Stigma: number analyzed (Participants) | 15 | 4
  Change at Week 106: Stigma | -0.1 (12.67) | 4.5 (10.25)
  Baseline: Behavior | 51.4 (10.39) | 45.8 (9.33)
  Change at Week 106: Behavior: number analyzed (Participants) | 15 | 4
  Change at Week 106: Behavior | 0.2 (5.92) | 7.3 (6.55)
  Baseline: General-health | 50.5 (10.02) | 49.0 (8.40)
  Change at Week 106: General health: number analyzed (Participants) | 15 | 4
  Change at Week 106: General health | -1.3 (10.98) | -2.0 (10.86)
  Baseline: Quality-of-life | 49.5 (9.71) | 50.7 (9.98)
  Change at Week 106: Quality-of-life: number analyzed (Participants) | 15 | 4
  Change at Week 106: Quality-of-life | 1.1 (9.46) | 3.3 (12.28)

ADVERSE EVENTS:
Time Frame: From Visit 1 up to 30 days after the last study visit, or until resolution, whichever came first (up to approximately Week 106)
Arm/Group | Rufinamide | Any Other Approved Antiepileptic Drug
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/12
Serious Adverse Events (participants affected / at risk) | 10/25 | 5/12
Other Adverse Events (participants affected / at risk) | 21/25 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rufinamide (N=25) | Any Other Approved Antiepileptic Drug (N=12)
Blindness (Eye disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1
Encephalitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized tonic-clonic seizure (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 3
Status epilepticus (Nervous system disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rufinamide (N=25) | Any Other Approved Antiepileptic Drug (N=12)
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 7 | 1
Gait disturbance (General disorders) | 2 | 1
Pyrexia (General disorders) | 4 | 3
Bronchiolitis (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
Otitis media (Infections and infestations) | 4 | 0
Pneumonia (Infections and infestations) | 4 | 0
Sinusitis (Infections and infestations) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 4
Blood bicarbonate decreased (Investigations) | 2 | 1
Weight decreased (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1
Somnolence (Nervous system disorders) | 5 | 0
Irritability (Psychiatric disorders) | 3 | 1
Sleep disorder (Psychiatric disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Circadian rhythm sleep disorder (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Strabismus correction (Surgical and medical procedures) | 0 | 1
Aggression (Psychiatric disorders) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No